CLINICAL TRIAL: NCT00621023
Title: A Pilot Phase II Study of Decitabine, Arsenic Trioxide and Ascorbic Acid for Patients With Myelodysplastic Syndrome
Brief Title: Cephalon Decitabine, Arsenic Trioxide and Ascorbic Acid for Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Cephalon (Industry); Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00011792; 7667A (Other: Cephalon)
Record Dates: First submitted 2007-12-26; First posted 2008-02-22 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic syndrome; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine; Arsenic Trioxide; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Drug: Decitabine, Arsenic Trioxide and Ascorbic Acid for MDS
  Interventions: Drug: Decitabine, Arsenic Trioxide and Ascorbic Acid

INTERVENTIONS:
Drug: Decitabine, Arsenic Trioxide and Ascorbic Acid — Subjects receive decitabine 20 mg/m2 IV over one hour for days1-5 of each cycle, and arsenic trioxide 0.25 mg/kg IV for days 1-5 of cycle 1 followed by 0.25 mg/kg twice weekly (Mon-Thursday or Tues-Fri) for all remaining cycles. Patients will have transfusion and supportive care therapy administered per the treating physician's discretion. Patients with a response after 4 cycles of therapy may choose to continue on two more cycles of decitabine with arsenic and ascorbic acid given only during the first week of those two additional cycles.
  Other Names: Decitabine, ATO

SUMMARY:
This will be an open-label, non-randomized trial pilot phase II trial open to patients with myelodysplastic syndrome. The purpose of the study is to find out if the combination of decitabine, arsenic trioxide and ascorbic acid is safe.

DETAILED DESCRIPTION:
Conventional therapy for MDS has been poor at best. Supportive care with transfusion therapy and antibiotics have remained an option for all patients with myelodysplastic syndrome (MDS).

The only known curative therapy is an allogeneic bone marrow transplant. However due to its high morbidity in this elderly population and the lack of available donors, it is estimated that less than 5% of patients with MDS are candidates for this type of aggressive therapy. Investigational therapies are thus warranted in MDS.

Decitabine shows significant clinical activity in patients with MDS, with moderate toxicity. The major toxicity is myelosuppression with subsequent infection occurring in 20-25% of patients.

Arsenic trioxide is an FDA approved drug for the treatment of patients with acute promyelocytic leukemia (APL) who are refractory to, or have relapsed from, retinoid and anthracycline chemotherapy. Two pivotal studies of arsenic trioxide in the setting of relapsed APL showed a complete remission rate of 87% with a 36 month survival estimate of 50%. As of May 2004, over 800 patients had received arsenic trioxide in clinical studies or through a compassionate use program, and an additional 3600 patients had received the drug in clinical practice.

Arsenic trioxide shows clinical activity in MDS. Side effects have been noted and are manageable.

Adult patients with an established diagnosis of MDS will receive decitabine 20 mg/m2 IV over one hour for days1-5 of each cycle, and arsenic trioxide 0.25 mg/kg IV for days 1-5 of cycle 1 followed by 0.25 mg/kg twice weekly (Mon-Thursday or Tues-Fri) for all remaining cycles. The dose of ascorbic acid will be 1000 mg in 100 mL a solution of 5% dextrose in water (D5W) (protected from light and air) administered as an IV infusion over 15 to 30 minutes and administered within 30 minutes after arsenic trioxide administration.

Each cycle will consist of 4 weeks of treatment, and patients will be assessed each cycle for toxicity, and after 4 cycles for response as defined by the International Working Group (IWG - see section 8.0). Patients will have transfusion and supportive care therapy administered per the treating physician's discretion.

Patients with a response (complete response - CR, partial remission - PR, or hematologic improvement) after 4 cycles of therapy may choose to continue on two more cycles of decitabine with arsenic and ascorbic acid given only during the first week of those two additional cycles.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of MDS (de novo or secondary) fitting either the French American British Cooperative Group (FAB) or World Health Organization (WHO) classification systems as determined by a complete blood count (CBC) and bone marrow biopsy. Patients with >20% bone marrow blasts but <30% bone marrow blasts who would be classified as refractory anemia with excess blasts (RAEB-t) in the FAB and acute myeloid leukemia (AML) in the WHO systems are still eligible for this study. Patients with low risk MDS (IPSS scores low or intermediate -1 (INT-1) must be transfusion dependent to be eligible. Transfusion dependent will be defined as having 2 or more transfusion events within a 90 day period.
* Eastern Oncology Cooperative Group (ECOG) or WHO performance status of 0-2 (Appendix)
* Able to provide written informed consent.

Exclusion Criteria:

* Pregnant females
* AML defined as > 30% bone marrow blasts.
* Any malignant disease within the past 2 years, except cervical carcinoma, basal cell carcinoma of the skin, and squamous cell carcinoma of the skin..
* Off all prior treatment for MDS for at least 4 weeks from entry.
* Off any investigational agents for at least 4 weeks from entry.
* Uncontrolled cardiac disease or congestive heart failure as defined by New York Heart Association criteria of Class III or greater.
* Uncontrolled pulmonary disease.
* Uncontrolled or active viral or bacterial infection. All infections must have been fully treated with antibiotics.
* HIV +
* Lab values as specified in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos de Castro, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period occurred from November 2007 to April 2010 at Duke University Medical Center.
Pre-assignment Details: 1 patient was consented and found to be ineligible, and did not participate in the study.
Groups:
- All Participants: Drug: Decitabine, Arsenic Trioxide and Ascorbic Acid for MDS
  Decitabine, Arsenic Trioxide and Ascorbic Acid : Subjects receive decitabine 20 mg/m2 IV over one hour for days1-5 of each cycle, and arsenic trioxide 0.25 mg/kg IV for days 1-5 of cycle 1 followed by 0.25 mg/kg twice weekly (Mon-Thursday or Tues-Fri) for all remaining cycles. Patients will have transfusion and supportive care therapy administered per the treating physician's discretion. Patients with a response after 4 cycles of therapy may choose to continue on two more cycles of decitabine with arsenic and ascorbic acid given only during the first week of those two additional cycles.
Period: Overall Study
Arm/Group | All Participants
Started | 6
Completed | 0 (Completed is defined as 5 years of follow up.)
Not Completed | 6
Not completed — Death | 5
Not completed — Follow up discontinued | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With an Overall Response of Complete Response (CR) or Partial Response (PR)
Description: Complete response and Partial response are defined using 2000 international working group (IWG) criteria. The Primary criteria for a CR is a repeat bone marrow showing < 5% myeloblasts with normal maturation of all cell lines, with no evidence for dysplasia . A PR meets all the CR criteria except Blasts decreased by >50% over pretreatment, or a less advanced myelodysplastic syndrome (MDS) French American British (FAB) classification than pretreatment.
Time Frame: after 4 cycles of therapy
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 6
participants | 0

2. Secondary Outcome: Duration of a Complete or Partial Response Based on Number of People Who Responded.
Description: Number of months a complete or partial response was maintained.
Time Frame: Up to 5 years or until death
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients With an Unacceptable Toxicity
Description: Any of the following non-hematologic toxicities that causes a patient's therapy to be suspended or discontinued: Creatinine > 2x baseline value; serum glutamate oxaloacetate transaminase (SGOT), serum glutamate pyruvate transaminase (SGPT), Total bilirubin > 2x the upper limit of normal; Febrile neutropenia; Uncontrolled infection; Hepatotoxicity defined as an increase in serum bilirubin, SGOT, or alkaline phosphatase to >5 times baseline value); nephrotoxicity (defined as serum creatinine >3.5 times the ULN); neurological impairment (defined as somnolence, seizures, or impaired mentation); severe peripheral neuropathy, or any non-hematologic grade 4 toxic event.
Time Frame: During the treatment period and for 30 days after last dose of study drug
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 6
participants | 4

ADVERSE EVENTS:
Time Frame: During the treatment period and 30 days after last dose of study drug.
Description: Adverse Events are included regardless of attribution to study drug
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=6)
Hematoma (Vascular disorders) | 1 (1)
Infection with Grade 3 or 4 neutrophils - lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with Grade 3 or 4 neutrophils - Urinary tract not otherwise specified (Infections and infestations) | 1 (1)
Infection with unknown ANC - urinary tract not otherwise specified (Infections and infestations) | 1 (1)
Pain - Cardiac/heart (Cardiac disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile neutropenia (fever of unknown origin without documented infection) (Blood and lymphatic system disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=6)
Hemoglobin (Blood and lymphatic system disorders) | 2 (5)
Leukocytes (total WBC) (Investigations) | 2 (9)
Neutrophils / granulocytes (ANC / AGC) (Investigations) | 2 (13)
Platelets (Investigations) | 2 (7)
Prolonged QTc interval (Investigations) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (7)
Insomnia (Psychiatric disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (3)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (1)
Weight gain (Investigations) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Heartburn / dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (6)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hemorrhage / Bleeding - Other (Vascular disorders) | 1 (1)
Petechiae / purpura (hemorrhage / bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 1 (2)
Edema: limb (General disorders) | 1 (1)
Edema: trunk/genital (General disorders) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (5)
Alkaline phosphatase (Investigations) | 1 (5)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (5)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 1 (4)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (5)
Creatinine (Investigations) | 1 (3)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (5)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (10)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (2)
Dizziness (Nervous system disorders) | 2 (4)
Mood Alteration - Anxiety (Psychiatric disorders) | 1 (1)
Mood Alteration - Depression (Psychiatric disorders) | 2 (2)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (2)
Pain - back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Chest / thorax NOS (General disorders) | 1 (1)
Pain - kidney (Renal and urinary disorders) | 1 (1)
Pain - other (General disorders) | 1 (3)
Pain - skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pain - stomach (Gastrointestinal disorders) | 1 (1)
Pain - urethra (Renal and urinary disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Voice changes / dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary frequency / urgency (Renal and urinary disorders) | 2 (2)
Infection with unknown ANC - urinary tract not otherwise specified (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment stopped early, which lead to a small number of subjects analyzed. The subjects who were enrolled did complete the entire protocol and their data was analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No